CLINICAL TRIAL: NCT03375242
Title: XALKORI ROS1+NSCLC DRUG USE INVESTIGATION
Brief Title: Safety and Efficacy of Xalkori ROS1
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A8081051; NCT03375242 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- crizotinib
  Interventions: Drug: crizotinib

INTERVENTIONS:
Drug: crizotinib — XALKORI® Capsule 200 mg／XALKORI® Capsule 250 mg Frequency and duration are according to Package Insert as follows. " The recommended dose schedule of crizotinib is 250 mg taken orally twice daily. Dosing interruption and/or dose reduction may be required based on patients' clinical status. "
  Other Names: XALKORI® Capsule 200 mg／XALKORI® Capsule 250 mg

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the LPD (unknown adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3)factors considered to affect the safety and/or efficacy of this drug.

ELIGIBILITY:
Inclusion Criteria:

* patients with unresectable progressive/recurrent NSCLC who are naive to XALKORI and whose tumor is ROS1 gene positive

Exclusion Criteria:

* Patients with past history of hypersensitivity to any of the ingredients of XALKORI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-10-25 (Actual); Primary Completion 2027-03-26 (Estimated); Study Completion 2027-03-26 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse drug reactions in this surveillance. | 52 weeks

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 12, 24, 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A8081051